CLINICAL TRIAL: NCT00762242
Title: Metabolomic Profiling of Novel Mediators of Vascular Function
Status: Terminated | Type: Observational
Why Stopped: Study enrollment was no adequate.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua A. Beckman, MD, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2007P-000669
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: metabolomics; flow-mediated vasodilation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples for assays of novel biomarkers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Blood sampling and brachial artery ultrasound
  Interventions: Procedure: blood sampling and brachial artery ultrasound

INTERVENTIONS:
Procedure: blood sampling and brachial artery ultrasound — Intravenous blood sampling will be performed before and 15 seconds, 30 seconds, 1,2,5,10,and 30 minutes following an ischemic stimulus (inflation of a blood pressure cuff to suprasystolic pressure for 5 minutes)
  Brachial artery ultrasound imaging will be performed before and 1 minute after a 5 minute ischemic stimulus, to assess endothelium-dependent vasodilation of the brachial artery.
  Following completion of blood sampling, an additional "resting" image of the brachial artery will be obtained. Sub-lingual nitroglycerin will be administered, and the artery will be imaged again after 3 minutes, to assess endothelium-independent vasodilation.

SUMMARY:
The purpose of this study is to identify and characterize specific chemicals and metabolic pathways that change with forearm ischemia. These changes will be compared with forearm blood flow and flow-mediated vasodilation of the brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Type 2 diabetes mellitus

Exclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetics taking insulin, thiazolidinediones (rosiglitazone or pioglitazone), an amylin analog (Symlin [pramlintide]), or incretin mimetics (Byetta [exenatide])
* Pregnancy
* Uncontrolled hypertension, > 180/100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
change from baseline (pre-forearm ischemia) in circulating metabolites compared with post-ischemic forearm measurements | pre/post 5 minute ischemic stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A. Beckman, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States